CLINICAL TRIAL: NCT00219180
Title: An 8-week Multi-center, Dose Escalation Study to Evaluate the Efficacy and Safety of Aliskiren (150 mg and 300 mg) Administered Alone and in Combination With Valsartan (160 mg and 320 mg) in Patients With Hypertension
Brief Title: Clinical Study to Evaluate Efficacy and Safety of Aliskiren (150mg & 300mg) Administered Alone and in Combo With Valsartan (160mg and 320mg) in Patients With High Blood Pressure
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CSPP100A2327
Record Dates: First submitted 2005-09-12; First posted 2005-09-22 (Estimated); Last update posted 2017-05-17 (Actual); Status verified 2017-05

CONDITIONS: Hypertension
Keywords: Hypertension, Aliskiren
MeSH Terms: conditions — Hypertension | interventions — aliskiren

INTERVENTIONS:
Drug: aliskiren

SUMMARY:
To evaluate the efficacy and safety of aliskiren alone and in combination with valsartan given to patients with essential hypertension

ELIGIBILITY:
Inclusion Criteria

* Patients with essential hypertension
* Patients who are eligible and able to participate in the study

Exclusion Criteria

* Severe hypertension
* History or evidence of a secondary form of hypertension
* History of Hypertensive encephalopathy or cerebrovascular accident

Other protocol-defined exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1797 (Actual)
Dates: Start 2005-06; Primary Completion 2006-09 (Actual); Study Completion 2006-09 (Actual)

PRIMARY OUTCOMES:
Change from baseline in diastolic blood pressure after week 8

SECONDARY OUTCOMES:
Change from baseline in systolic blood pressure after week 8
Diastolic blood pressure < 90 mmHg or a reduction of > 10 mmHg after 4 and 8 weeks
Blood pressure control target of < 140/90 mmHg after 4 and 8 weeks
Evaluate 24-hour ambulatory blood pressure monitoring in a subset of patients

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (2):
- Novartis Pharmaceuticals, East Hanover, New Jersey, United States
- Investigative Centers, Germany

REFERENCES:
- [Derived] Wang GM, Li LJ, Fan L, Xu M, Tang WL, Wright JM. Renin inhibitors versus angiotensin receptor blockers for primary hypertension. Cochrane Database Syst Rev. 2025 Feb 27;2(2):CD012570. doi: 10.1002/14651858.CD012570.pub2. PMID 40013543
- [Derived] Oparil S, Yarows SA, Patel S, Fang H, Zhang J, Satlin A. Efficacy and safety of combined use of aliskiren and valsartan in patients with hypertension: a randomised, double-blind trial. Lancet. 2007 Jul 21;370(9583):221-229. doi: 10.1016/S0140-6736(07)61124-6. PMID 17658393